CLINICAL TRIAL: NCT07228468
Title: Home-Based Transcranial Direct Current Stimulation in Major Depressive Disorder: a Multi-Centre, Two-Parallel Group, Superiority Randomised Controlled Trial
Brief Title: Home-Based Transcranial Direct Current Stimulation In Major Depressive Disorder (HOME)
Acronym: HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government); Cardiff and Vale University Health Board (Other Government); Northumberland, Tyne and Wear NHS Foundation Trust (Other); Northamptonshire Healthcare NHS Foundation Trust (Other); South London and Maudsley NHS Foundation Trust (Other); Southern Health NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIHR165425; NIHR165425 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: transcranial direct current stimulation; tDCS; major depression; MDD; major depressive disorder; brain stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive active transcranial direct current stimulation (tDCS) OR treatment as usual (TAU).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (No Intervention): Treatment as usual will consist of standard care, such as psychotherapy and/or antidepressant medication or no treatment, as decided by participant and treating clinician.
- transcranial direct current stimulation + treatment as usual (tDCS + TAU) (Experimental): In addition to receiving treatment as usual, participants randomized to receive tDCS will engage in a 10-week treatment protocol of active tDCS which participants will administer at home. Stimulation schedule is 5 sessions per week for 3 weeks followed by 3 sessions per week for 7 weeks, for a total of 36 sessions in 10 weeks. tDCS device is headset with bifrontal montage, anode at left dorsolateral prefrontal cortex (DLPFC) and cathode at right DLPFC (EEG positions F3 and F4, respectively). Stimulation is 2 mA for 30 minutes with a gradual ramp up over 30 seconds. Electrode area is 23 cm2.
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Participants randomised to the tDCS treatment arm will use a tDCS device which is a headset with the anode positioned over left dorsolateral prefrontal cortex (DLPFC) and cathode over right DLPFC (EEG positions F3 and F4, respectively). Treatment protocol consists of 5 tDCS sessions per week for 3 weeks followed by 3 tDCS sessions per week for 7 weeks, for a total of 36 sessions in 10 weeks. tDCS stimulation is 2 mA for 30 minutes with gradual ramp up over 30 seconds at the start and end of each session.
  Arms: transcranial direct current stimulation + treatment as usual (tDCS + TAU)

SUMMARY:
Depression is a prevalent and debilitating disorder. The most common treatments are antidepressant medications and talking therapies. However, for many individuals, these are not their treatment of choice. Furthermore, even following a full course of treatment with an antidepressant or talking therapy, over one third of patients continue to be unwell.

The novel brain stimulation treatment, transcranial direct current stimulation (tDCS), is a potential first-line treatment for major depression. The present research question is whether home-based tDCS is an effective treatment for major depression for adults with major depression.

Participants will be randomised to receive either a 10-week course of active tDCS treatment in addition to their standard care (Treatment as Usual), or to only receive Treatment as Usual. Participants will be followed up for 6-months after the start of the treatment began.

After the 6-month follow-up visit, all participants from both groups can choose to continue/start the tDCS treatment. There will be a final follow-up visit 3 months later (9 months from the original treatment start of the trial).

DETAILED DESCRIPTION:
Current pharmacotherapy and psychotherapy treatments for major depressive disorder (MDD) often fall short in efficacy and patient satisfaction, highlighting a critical need for innovative, effective and acceptable treatment options. Transcranial direct current stimulation (tDCS) has emerged as a promising treatment, offering a non-invasive method to modulate brain activity and alleviate depressive symptoms that can be provided at home.

This trial builds on our work and aims to evaluate the effectiveness and cost-effectiveness of home-based tDCS as a treatment for MDD in the NHS. The trial is a multi-centre pragmatic RCT to evaluate the real-life clinical effectiveness and cost-effectiveness of tDCS combined with treatment as usual (TAU) as compared to TAU alone following a 10-week treatment period and at a 6-month follow up. Depressive symptoms will be measured by the clinician-rated Montgomery-Åsberg Depression Rating Scale (MADRS). We will further assess impact on self-report depressive symptoms, anxiety symptoms, remission, acceptability and quality of life. We will conduct in-depth process evaluation, economic evaluation, and implementation work to investigate operational challenges of integrating home-based tDCS into existing NHS care pathways and to inform scalability in primary care settings.

438 Participants will be aged 18 years or over, diagnosed with MDD with at least moderate severity of depressive symptoms and medication free or taking stable antidepressant medication or in psychotherapy for at least 6 weeks before enrolment. Participants will be randomly assigned in a 1:1 ratio to either TAU or TAU+tDCS.

Participants randomised to the TAU treatment arm will continue with standard care including psychotherapy and/or antidepressant medication, as decided by participant and treating clinician. Participants randomised to the tDCS treatment arm will use a tDCS device which is a headset with the anode positioned over left dorsolateral prefrontal cortex (DLPFC) and cathode over right DLPFC (EEG positions F3 and F4, respectively). Treatment protocol consists of 5 tDCS sessions per week for 3 weeks followed by 3 tDCS sessions per week for 7 weeks, for a total of 36 sessions in 10 weeks. tDCS stimulation is 2 mA for 30 minutes with gradual ramp up over 30 seconds at the start and end of each session.

The primary outcome is the difference in depressive symptoms between treatment arms at 10-week end of treatment as measured by MADRS and the key secondary outcome is the long term clinical effectiveness as measured by difference in depressive symptoms between treatment arms at 6-month follow up as measured by MADRS.

After the 6-month follow up, a 3-month extension follow up phase will give all participants the opportunity to use the tDCS device.

This research addresses an unmet need for new treatment options for MDD, thereby benefiting people with MDD, improving NHS care pathways, and expanding scientific knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or over
2. Current episode of depression based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria (APA, 2013) for major depressive disorder (MDD) as assessed by structured clinical assessment, Mini-International Neuropsychiatric Interview (MINI) (Sheehan et al., 1998)
3. Having at least a moderate severity of depressive symptoms as measured by a score of at least 18 in MADRS
4. Either not taking antidepressant medication or taking a stable dose of antidepressant medication for at least 6 weeks before enrolment.
5. Either not currently in psychotherapy or in ongoing psychotherapy for at least 6 weeks before enrolment.
6. Being under the care of GP
7. Agreeable for GP to be regularly informed about study participation
8. Able to provide written, informed consent

Exclusion Criteria:

1. Significant suicide risk as measured by answering 'yes' to questions 4, 5 or 6 on the Columbia Suicide Severity Rating Scale (C-SSRS) Screen (Posner et al., 2011)
2. Primary comorbid psychiatric disorder (e.g. obsessive compulsive disorder) based on DSM-5 criteria as assessed in MINI
3. Current daily use of medications that affect cortical excitability (e.g. benzodiazepines)
4. Current illicit drug use or heavy alcohol use with high risk of alcohol use disorder as measured by a score of 8 or more in Alcohol use disorders identification test consumption (AUDIT C) (Khadjesari et al., 2017; NICE, 2023)
5. History of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), cranial electrotherapy stimulation (CES), transcranial direct current stimulation (tDCS), deep brain stimulation (DBS), or other brain stimulation
6. History of esketamine / ketamine for treatment of depression
7. History of psychosurgery for depression
8. Having cognitive impairment (e.g. dementia)
9. Current medical disorder or neurological disorder that may mimic mood disorder (e.g. hormonal disorder, unstable heart disease)
10. Have any implant in the brain or neurocranial defect
11. Have shrapnel or any ferromagnetic material in the head
12. Have any active implantable medical device (e.g. pacemaker)
13. If female and of child-bearing potential, currently pregnant or planning to become pregnant during the study
14. Concurrent enrolment in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 10 weeks
  To evaluate tDCS clinical effectiveness as the difference in depressive symptom severity at end of 10-week treatment period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 months
  To evaluate tDCS clinical effectiveness as the difference in depressive symptom severity at end of 6 month follow-up period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Hamilton Depression Rating Scale (HDRS) | 10 weeks
  To evaluate tDCS clinical effectiveness as the difference in depressive symptom severity at end of 10-week treatment period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Hamilton Anxiety Rating Scale (HAMA) | 10 weeks
  To evaluate tDCS clinical effectiveness as the difference in anxiety symptom severity at end of 10-week treatment period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Montgomery-Åsberg Depression Rating Scale-Self Report (MADRS-S) | 10 weeks
  To evaluate tDCS clinical effectiveness as the difference in depressive symptom severity at end of 10-week treatment period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Hamilton Depression Rating Scale (HDRS) | 6 months
  To evaluate tDCS clinical effectiveness as the difference in depressive symptom severity at end of the 6 month follow-up period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Hamilton Anxiety Rating Scale (HAMA) | 6 months
  To evaluate tDCS clinical effectiveness as the difference in anxiety symptom severity at end of the 6 month follow-up period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Montgomery-Åsberg Depression Rating Scale-Self Report (MADRS-S) | 6 months
  To evaluate tDCS clinical effectiveness as the difference in depressive symptom severity at end of the 6 month follow-up period between two treatment arms: those receiving treatment as usual (TAU) alone and those receiving TAU plus tDCS
Montgomery-Åsberg Depression Rating Scale (MADRS) clinical response | 10 weeks
  To evaluate treatment response at the 10-week end of treatment period between treatment arms. Treatment response is defined as an improvement of 50% or more from baseline MADRS score.
Montgomery-Åsberg Depression Rating Scale (MADRS) treatment remission | 10 weeks
  To evaluate treatment remission at the 10-week end of treatment period between treatment arms. Treatment remission is defined as a MADRS score of 10 or less.
Montgomery-Åsberg Depression Rating Scale (MADRS) clinical response | 6 months
  To evaluate treatment response at the 6 month end of follow-up period between treatment arms. Treatment response is defined as an improvement of 50% or more from baseline MADRS score.
Montgomery-Åsberg Depression Rating Scale (MADRS) treatment remission | 6 months
  To evaluate treatment remission at the 6 month follow-up period between treatment arms. Treatment remission is defined as a MADRS score of 10 or less.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Fu, MD, PhD, Principal Investigator — King's College London
Locations (6):
- United Kingdom (6):
  - Cardiff and Vale Health Board, Cardiff
  - South London and Maudsley NHS Foundation Trust, London
  - Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle
  - Northamptonshire Healthcare NHS Foundation Trust, Northampton
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham
  - Hampshire and Isle of Wight Healthcare NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on request.
Supporting Information: Study Protocol, SAP
Time Frame: a maximum of 1 year after publication of study results
Access Criteria: Individual access by request